CLINICAL TRIAL: NCT04668352
Title: A Phase 3 Study to Determine if RTB101 Prevents Clinically Symptomatic Respiratory Illness in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Restorbio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RTB-101-204
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — dactolisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dactolisib 10mg once daily (Experimental)
  Interventions: Drug: Dactolisib
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dactolisib — TORC1 inhibitor
  Arms: Dactolisib 10mg once daily
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To determine if RTB101 as compared to placebo decreases the percentage of subjects with clinically symptomatic respiratory illness (with or without an associated laboratory-confirmed pathogen) through Week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male and female subjects who, in the clinical judgement of the Investigator, are without unstable medical conditions defined as conditions that require acute medical intervention or ongoing adjustments of concomitant medications (as determined by medical history, current concomitant medications and laboratory test results at Screening, and physical examination, electrocardiogram (ECG) and vital signs at Screening and Baseline).
3. Subjects must be ≥65 years of age.
4. Subjects should require no or minimal assistance with self-care and activities of daily living. Subjects in assisted-living or long-term care residential facilities that provide minimal assistance are eligible.
5. Females must be post-menopausal. Women are considered postmenopausal and not of childbearing potential if they have had:

   * 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) OR
   * Surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks prior to Screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment will she be considered not of childbearing potential.
6. Sexually active male subjects with a partner of child-bearing potential must be willing to wear a condom while on study drug and for 1 week after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men with a partner of child-bearing potential to prevent delivery of the drug via seminal fluid.
7. Subject must weigh at least 40 kg.
8. Subject must be able to communicate well with the Investigator, and to understand and comply with the requirements of the study including completing a daily eDiary at home.

Exclusion Criteria:

1. Any subject who:

   * Is a current smoker as assessed by medical history or a positive serum cotinine test (or positive urine cotinine test if serum cotinine testing is unavailable) at Screening. Stopped smoking ≤1 year prior to Screening.
   * Is a previous smoker with a ≥10 pack year smoking history. Has a household member who currently smokes in the house
2. Subjects with a medical history of clinically significant lung diseases other than asthma (e.g., chronic obstructive pulmonary disease (COPD), emphysema, interstitial pulmonary fibrosis (IPF), bronchiectasis, etc.).
3. Subjects with a Mini Mental Status Examination (MMSE) score <24 at Screening.
4. Subjects with current evidence of a serious and/or unstable medical disorder including cardiovascular, respiratory, gastrointestinal, renal (including subjects with an estimated glomerular filtration rate (eGFR) as estimated by the modified diet in renal disease (MDRD) GFR equation that is ≤30 mL/min/1.73m2), or hematologic disorders.
5. The following cardiac conditions:

   * Unstable angina pectoris or acute ischemic changes on ECG at Screening or Baseline
   * History of myocardial infarction (MI), coronary bypass surgery, or any percutaneous coronary intervention (PCI) within 6 months prior to Screening
   * New York Heart Association functional classification IIIIV congestive heart failure
   * Unstable or life-threatening cardiac arrhythmia, chronic stable atrial fibrillation is allowed.
   * QTcF>480 msec at Screening or Baseline
6. Subjects with history of malignancy in any organ system within the past 5 years, EXCEPT for the following:

   * Localized basal cell or squamous cell carcinoma of the skin.
   * Prostate cancer confined to the gland (AJCC stage T2N0M0 or better).
   * Cervical carcinoma in situ.
   * Breast cancer localized to the breast.
7. Any RTI or acute significant illness (based on the subject's medical history and the clinical judgement of the Investigator) which has not resolved at least two (2) weeks prior to Baseline.
8. Subjects with a history of systemic autoimmune diseases (e.g., lupus, inflammatory bowel disease, rheumatoid arthritis, etc.), or receiving immunosuppressive therapy (such as mycophenolate, tacrolimus, cyclosporine, azathioprine, infliximab) including chronic use of prednisone >10 mg daily (however, inhaled corticosteroids and the acute use of higher doses of prednisone to treat conditions such as exacerbation of asthma or other acute conditions are allowed).
9. Subjects with Type I diabetes mellitus.
10. Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further evaluation.
11. Subjects with any one of the following during Screening:

    * white blood cell (WBC) count <2.0 x103/microL.
    * neutrophil count <1.0 x 103/microL.
    * platelet count <75 x 103/microL..
12. Subjects with a history of alcohol or drug abuse within 2 years of the Screening visit.
13. Subjects with any conditions affecting absorption, distribution, or metabolism of the study drug (e.g., inflammatory bowel disease, gastric or duodenal ulcers, or hepatic disease). For subjects with biochemical evidence of liver injury as indicated by abnormal liver function tests:

    * Any single parameter of alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase or serum bilirubin must not exceed 1.5 x upper limit of normal (ULN) in subjects who do not have Gilbert's syndrome. If the subject has a history of Gilbert's syndrome, direct and indirect reacting bilirubin should be differentiated, and the direct bilirubin must be less than 1.5 x ULN.
    * Any elevation above ULN of more than one parameter of ALT, AST, alkaline phosphatase or serum bilirubin will exclude a subject from participation in the study.
14. Subjects with a history of immunodeficiency diseases, including a positive human immunodeficiency virus (HIV) test result.
15. Infection with Hepatitis B virus (HBV) or Hepatitis C virus (HCV).
16. Subjects who require treatment with strong CYP3A4 or CYP1A2 inhibitors or inducers, or subjects who require treatment with digoxin.
17. Use of any other investigational medication or participation in any other investigational study within 5 half-lives of the investigational medication, or within 30 days, whichever is longer; or longer if required by local regulations.
18. Subjects who have received an organ transplant.
19. Subjects who previously received treatment with RTB101 in another clinical study (e.g., CBEZ235Y2201, RTB-BEZ235-202, or RTB-101-203).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Quinn, MD, Principal Investigator — P3 Research Ltd.
Locations (1):
- P3 Research Ltd., Wellington, New Zealand

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Dactolisib 10mg Once Daily
Started | 511 | 513
Completed | 510 | 511
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dactolisib 10mg Once Daily | Total
Number analyzed (Participants) | 510 | 511 | 1021
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (5.83) | 72.6 (5.81) | 72.8 (5.82)
Age, Customized [Count of Participants; unit: Participants]
  >=65 and <85 years | 486 | 488 | 974
  >=85 years | 24 | 23 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286 | 292 | 578
  Male | 224 | 219 | 443
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 503 | 510 | 1013
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 9 | 13
  Native Hawaiian or Other Pacific Islander | 8 | 11 | 19
  Black or African American | 0 | 0 | 0
  White | 498 | 490 | 988
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 510 | 511 | 1021
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (5.13) | 29.2 (5.47) | 29.0 (5.31)
Received Current Season Influenza Vaccination [Count of Participants; unit: Participants] | 407 | 415 | 822

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Clinically Symptomatic Respiratory Illness
Description: To determine if RTB101 as compared to placebo decreases the percentage of subjects with clinically symptomatic respiratory illness (with or without an associated laboratory-confirmed pathogen) through Week 16
Time Frame: Week 0-16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dactolisib 10mg Once Daily
Number analyzed (Participants) | 510 | 511
Participants | 125 | 134

ADVERSE EVENTS:
Time Frame: Up to Week 16
Arm/Group | Placebo | Dactolisib 10mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/510 | 1/511
Serious Adverse Events (participants affected / at risk) | 32/510 | 31/511
Other Adverse Events (participants affected / at risk) | 371/510 | 386/511
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=510) | Dactolisib 10mg Once Daily (N=511)
Splenic embolism (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Coronary artery dissection (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Metabolism and nutrition disorders (Investigations) | 1 | 0
Hyponatraemia (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal embolism (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Cancer surgery (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=510) | Dactolisib 10mg Once Daily (N=511)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Splenic embolism (Blood and lymphatic system disorders) | 1 | 3
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 19 | 16
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 10 | 6
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery dissection (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 4 | 4
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 2 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 3
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 2
Meniere's disease (Ear and labyrinth disorders) | 1 | 1
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 3
Hypothyroidism (Endocrine disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 1
Blepharitis (Eye disorders) | 2 | 1
Cataract (Eye disorders) | 1 | 2
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 0 | 2
Episcleritis (Eye disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Eyelid haematoma (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Keratoconus (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 2 | 0
Macular degeneration (Eye disorders) | 1 | 0
Myopia (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0
Scleritis (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 1
Vitreous detachment (Eye disorders) | 0 | 2
Vitreous floaters (Eye disorders) | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 3
Change of bowel habit (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 6
Dental caries (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 34 | 35
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Discoloured vomit (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 2 | 1
Faeces hard (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 3 | 3
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 5
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 1
Lip ulceration (Gastrointestinal disorders) | 2 | 6
Mouth ulceration (Gastrointestinal disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 11 | 7
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 3
Tongue disorder (Gastrointestinal disorders) | 2 | 0
Tongue erythema (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 5
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Uvulitis (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 4
Adverse drug reaction (General disorders) | 0 | 1
Application site erosion (General disorders) | 0 | 1
Application site rash (General disorders) | 0 | 1
Asthenia (General disorders) | 7 | 9
Chest discomfort (General disorders) | 3 | 0
Chest pain (General disorders) | 6 | 5
Chills (General disorders) | 1 | 4
Drug intolerance (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 11 | 12
Influenza like illness (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Medical device pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 3 | 4
Pain (General disorders) | 8 | 5
Peripheral swelling (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 1
Therapeutic response unexpected (General disorders) | 59 | 66
Vessel puncture site bruise (General disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Allergy to plants (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 9 | 2
Abscess limb (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Anal candidiasis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteriuria (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 5
Bursitis infective (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Conjunctivitis (Infections and infestations) | 1 | 5
Corona virus infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 4
Ear infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 2 | 3
Furuncle (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 9 | 9
Gastroenteritis viral (Infections and infestations) | 1 | 1
Genital herpes (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 0 | 1
Infected bite (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Lice infestation (Infections and infestations) | 1 | 0
Lip infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 4 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Medical device site infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 0 | 1
Nasal herpes (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 1 | 2
Oral herpes (Infections and infestations) | 16 | 7
Otitis externa (Infections and infestations) | 4 | 4
Otitis media (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 1 | 1
Periodontitis (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 5 | 2
Root canal infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 6
Skin infection (Infections and infestations) | 0 | 5
Staphylococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 2
Tooth abscess (Infections and infestations) | 4 | 0
Tooth infection (Infections and infestations) | 2 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 21 | 15
Urosepsis (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 3 | 2
Viral rash (Infections and infestations) | 1 | 0
Viral rhinitis (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 2
Wound infection (Infections and infestations) | 2 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 1
Anal injury (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 2 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 3
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 2 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 10 | 22
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0
Dental restoration failure (Injury, poisoning and procedural complications) | 2 | 1
Extra dose administered (Injury, poisoning and procedural complications) | 1 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 28 | 20
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 3 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 3 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 7 | 10
Limb injury (Injury, poisoning and procedural complications) | 1 | 2
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 10 | 16
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 1
Nail injury (Injury, poisoning and procedural complications) | 0 | 1
Palate injury (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pharyngeal injury (Injury, poisoning and procedural complications) | 1 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural constipation (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 5 | 3
Repetitive strain injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 2 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 14 | 21
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 8 | 11
Skin wound (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 2 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 3 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 2
Alanine aminotransferase increased (Investigations) | 2 | 2
Biopsy skin (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood potassium increased (Investigations) | 0 | 5
Blood pressure increased (Investigations) | 2 | 3
Cardiac murmur (Investigations) | 3 | 2
Electrocardiogram QT prolonged (Investigations) | 3 | 7
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 1 | 0
Faecal volume increased (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 2 | 3
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Haematocrit increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 5
Hepatic enzyme increased (Investigations) | 0 | 1
Laboratory test abnormal (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1
Liver function test increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Occult blood positive (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 2 | 0
Red blood cells urine positive (Investigations) | 0 | 1
Renal function test abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 2
Urinary sediment present (Investigations) | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 1
Vitamin B12 decreased (Investigations) | 1 | 0
Vitamin D decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 2 | 1
White blood cell count increased (Investigations) | 1 | 0
White blood cells urine positive (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Salt craving (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 4
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 21
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 11
Bursitis (Musculoskeletal and connective tissue disorders) | 5 | 4
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 9
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 6
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 6
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 13
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Amnesia (Nervous system disorders) | 2 | 0
Aphonia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Circadian rhythm sleep disorder (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 13 | 13
Dizziness postural (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Facial neuralgia (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 26 | 37
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hyposmia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 6 | 9
Mental impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 2 | 2
Migraine with aura (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 2
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 4 | 3
Presyncope (Nervous system disorders) | 2 | 3
Sciatica (Nervous system disorders) | 2 | 1
Sedation (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 5 | 0
Tension headache (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Vascular parkinsonism (Nervous system disorders) | 1 | 0
Device breakage (Product Issues) | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 4
Apathy (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 4 | 3
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 1
Renal cyst (Renal and urinary disorders) | 0 | 2
Renal embolism (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 5 | 4
Renal infarct (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary tract discomfort (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 12 | 18
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal mucosal erosion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinitis perennial (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 8 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 5 | 6
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 2
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Onychomalacia (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 2
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 13
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 8 | 5
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Cancer surgery (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 2
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 1
Eyelid operation (Surgical and medical procedures) | 1 | 0
Gastric polypectomy (Surgical and medical procedures) | 1 | 0
Hernia repair (Surgical and medical procedures) | 0 | 1
Joint irrigation (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Lipoma excision (Surgical and medical procedures) | 1 | 0
Prostatectomy (Surgical and medical procedures) | 0 | 1
Ptosis repair (Surgical and medical procedures) | 0 | 1
Skin lesion removal (Surgical and medical procedures) | 2 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 2
Spinal decompression (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 2 | 1
Urethral dilation procedure (Surgical and medical procedures) | 1 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 3 | 5
Hot flush (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 9 | 19
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT04668352/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT04668352/SAP_001.pdf